CLINICAL TRIAL: NCT04288219
Title: Non-Invasive Positive Pressure Ventilation Management of High Altitude Pulmonary Edema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Himalayan Rescue Association (Unknown)
Responsible Party: Principal Investigator, N. Stuart Harris MD MFA, Chief, Division of Wilderness Medicine, Principal Investigator, Clinical Innstructor, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P003234
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: High Altitude Pulmonary Edema; Non-Invasive Positive Pressure Ventilation; Hypoxia
MeSH Terms: conditions — Altitude Sickness; Hypoxia | interventions — Nifedipine

STUDY DESIGN:
Masking Description: No masking will be done, as the CPAP device will be visible to both participants and investigators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Treatment (Active Comparator): Continuous supplemental oxygen and nifedipine 30mg will be administered to patients.
  Interventions: Drug: Nifedipine; Other: supplemental oxygen
- Non-Invasive Positive Pressure Ventilation Management (Experimental): CPAP at 10mmHg with supplemental oxygen, as well as nifedipine 30mg will be administered to patients.
  Interventions: Device: Non-Invasive Positive Pressure Ventilation; Drug: Nifedipine

INTERVENTIONS:
Device: Non-Invasive Positive Pressure Ventilation — Continuous positive airway pressure delivered by face mask at 10cmH2O
  Other Names: CPAP
  Arms: Non-Invasive Positive Pressure Ventilation Management
Drug: Nifedipine — Nifedipine 30mg, Pharmacotherapy
Other: supplemental oxygen — supplemental oxygen
  Arms: Standard of Care Treatment

SUMMARY:
Trial of Non-Invasive Positive Pressure Ventilation Management of High Altitude Pulmonary Edema

DETAILED DESCRIPTION:
Patients in the Everest area will assessed for evidence of acute HAPE. Subjects will be randomized and assigned to standard care options or treatment with Non-Invasive Positive Pressure Ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (age 18-80)
* Travel through Pheriche, Nepal
* Diagnosis of HAPE by symptoms, vital signs, and lung ultrasound

Exclusion Criteria:

* History of chronic respiratory conditions (asthma, COPD, ILD)
* Concomitant pneumonia or aspiration, cardiomyopathy, congestive heart failure
* Kidney disease
* Neurologic disorder
* Cognitive disorder
* Temporary altered mental status
* Use of phosphodiesterase inhibitors or nifedipine prior to diagnosis of HAPE
* Age under 18 or over 80
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Oxygen saturation | Up to 4 hours
  Displayed on pulse oximeter

SECONDARY OUTCOMES:
Ultrasonographic assessment of pulmonary edema | Up to 4 hours
  Quantification of B-lines
Subjective rating of dyspnea | Up to 4 hours
  Based on Dypnea Severity Scale (DSS)

CONTACTS AND LOCATIONS:
Locations (1):
- Himalayan Rescue Association, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No